CLINICAL TRIAL: NCT01730222
Title: A Phase I-II Study of PAXG in Stage III-IV Pancreatic Adenocarcinoma
Acronym: PACT-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACT-19; 2012-001763-75 (EudraCT Number)
Record Dates: First submitted 2012-11-04; First posted 2012-11-21 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic adenocarcinoma; stage III disease; stage IV disease; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Disease | interventions — Cisplatin; Capecitabine; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAXG regimen (Experimental): cisplatin at 30 mg/m2 on days 1 and 15, nab-paclitaxel at the RP2D on days 1 and 15, capecitabine at 1250 mg/ m2 days 1-28, gemcitabine at 800 mg/ m2 on days 1 and 15 every 4 weeks
  Interventions: Drug: cisplatin; Drug: capecitabine; Drug: gemcitabine; Drug: nab-paclitaxel
- gemcitabine + nab-paclitaxel (Active Comparator): gemcitabine at 1000 mg/ m2 on days 1, 8 and 15 every 4 weeks + nab-paclitaxel at 125 mg/ m2 on days 1, 8 and 15 every 4 weeks
  Interventions: Drug: gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: cisplatin — cisplatin at 30 mg/m2 on days 1 and 15
  Other Names: cisplatino TEVA
  Arms: PAXG regimen
Drug: capecitabine — capecitabine at 1250 mg/ m2 days 1-28
  Other Names: XELODA
  Arms: PAXG regimen
Drug: gemcitabine — gemcitabine at 800 mg/ m2 on days 1 and 15 in arm A; at 1000 mg/m2 on days 1, 8 and 15 in arm B
  Other Names: Gemzar
Drug: nab-paclitaxel — nab-paclitaxel at the recommended phase II dose day 1 and 15 in arm A; at 125 mg/m2 on days 1, 8 and 15 in arm B
  Other Names: abraxane

SUMMARY:
Four-drug combo yielded a statistically significant improvement in progression-free survival and overall survival compared to gemcitabine in patients with advanced pancreatic adenocarcinoma. Nab-Paclitaxel showed promising antitumor activity in patients with pancreatic cancer. Given the synergism of taxanes with gemcitabine, fluoropyrimidines and platinating agents the role of nab-Paclitaxel in a 4-drug regimen will be explored.

The aim of this trial is to determine the recommended dose of nab-paclitaxel in combination with cisplatin, capecitabine, and gemcitabine, PAXG regimen (Phase I), and to evaluate the feasibility and the activity of the PAXG regimen in patients with stage III and IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: PHASE I: to determine the recommended phase 2 dose of nab-paclitaxel in combination with cisplatin, capecitabine, and gemcitabine.

PHASE II: to evaluate the feasibility and the activity of the PAXG regimen in terms of 6-months progression-free survival in patients with stage III and IV pancreatic cancer.

OUTLINE Phase I - dose finding single institution trial, followed by a randomized open label multicenter phase II trial.

Phase II: Patients will be stratified by stage (III vs IV) and CA19.9 level (< 10 x ULN versus >10 x ULN); Patients will be randomly assigned to receive PAXG (arm A) or gemcitabine-nab-paclitaxel regimen (arm B).

Treatment plan (phase II):

Arm A: PAXG every 4 weeks (1 cycle): cisplatin at 30 mg/m2 on days 1 and 15, nab-paclitaxel at the RP2D on days 1 and 15, capecitabine at 1250 mg/ m2 days 1-28, gemcitabine at 800 mg/ m2 on days 1 and 15.

Arm B: Gemcitabine + nab-paclitaxel every 4 weeks (1 cycle): gemcitabine at 1000 mg/m2 on days 1, 8 and 15; nab-paclitaxel at 125 mg/mq on days 1, 8 and 15.

Treatment will be administered for a maximum of 6 cycles or until there is a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of pancreatic adenocarcinoma
* Stage III or IV disease
* Age > 17 < 76 years
* Karnofsky Performance Status > 50
* Measurable disease (only for phase II part)
* Adequate bone marrow (GB > 3500/mm3, neutrophils > 1500/mm3; platelets > 100000/mm3; hemoglobin > 10 g/dl), liver (total bilirubin < 2 mg/dL; SGOT e SGPT < 3 UNL) and kidney function (serum creatinin < 1.5 mg/dL;)
* Written informed consent

Exclusion Criteria:

* previous chemotherapy
* concurrent treatment with other experimental drugs
* previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin and of other neoplasms without evidence of disease at least from 5 years
* symptomatic brain metastases
* history of interstitial lung disease
* presence of serious disease which can compromise safety (cardiac failure, previous myocardial infarction within the prior 6 months, cardiac arrhythmia, history of psychiatric disabilities)
* pregnancy and lactating
* History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-11; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
first cycle toxicity for phase I part | after one month from treatment start
  Dose Limiting Toxicity definition: DLT will be defined as any of the following events attributable to the administered study drugs:
  * Hematologic toxicity
    * Grade ≥ 4 neutropenia lasting 7 days or more
    * Grade ≥ 3 febrile neutropenia or fever of unknown origin ≥ 38.5°C
    * Grade 4 thrombocytopenia
    * Grade 3 thrombocytopenia which required transfusions
  * Nausea or vomiting Grade ≥ 3 nausea or vomiting despite maximal antiemetic therapy
  * Diarrhea Grade ≥ 3 diarrhea despite optimal management of the event
  * Neurological toxicity Any Grade ≥ 2 neurological toxicity
  * Other non-hematologic toxicity Any grade ≥ 3 toxicities or representing a shift by 2 grades from baseline (in case of abnormal baseline)
  * Failure to recover Failure to recover to grade ≤ 1 toxicity (except alopecia) or to baseline values after delaying the initiation of next cycle by > 2 weeks.
progression-free survival for phase II part, stage IV patients | after 6 months from randomization
  rate of progression-free patients at 6 months from randomization
resectability rate for phase II part, stage III patients | after 4 and 6 months from treatment start
  rate of resectable patients at at time of CT evaluation and multidisciplinary assessment after 4 and 6 months from treatment start

SECONDARY OUTCOMES:
response rate | every two months up to 6 months during treatment; every 2-3 months afterwards until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  contrast enhanced CT scan tumor assessment
biochemical response rate | every month up to 6 months during treatment; every 2-3 months afterwards until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  blood sample for CA19.9 assessment
toxicity | every two weeks up to 26 weeks during treatment
  outpatients visits; laboratory
overall survival | From date of trial enrolment until the date of death from any cause, assessed every two weeks up to 26 weeks during treatment; every 2-3 months afterwards up to 60 months
  outpatients visit; phone interviews
Progression-free survival | From date of trial enrolment until the date of documented progression or date of death from any cause, whichever came first, assessed every two months up to 6 months during treatment; every 2-3 months afterwards up to 60 months
  contrast enhanced CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — IRCCS S RAFFAELE
Locations (1):
- IRCCS S Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reni M, Zanon S, Peretti U, Chiaravalli M, Barone D, Pircher C, Balzano G, Macchini M, Romi S, Gritti E, Mazza E, Nicoletti R, Doglioni C, Falconi M, Gianni L. Nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in metastatic pancreatic adenocarcinoma (PACT-19): a randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):691-697. doi: 10.1016/S2468-1253(18)30196-1. Epub 2018 Jul 7. PMID 30220407
- [Derived] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366
- [Derived] Reni M, Balzano G, Zanon S, Passoni P, Nicoletti R, Arcidiacono PG, Pepe G, Doglioni C, Fugazza C, Ceraulo D, Falconi M, Gianni L. Phase 1B trial of Nab-paclitaxel plus gemcitabine, capecitabine, and cisplatin (PAXG regimen) in patients with unresectable or borderline resectable pancreatic adenocarcinoma. Br J Cancer. 2016 Jul 26;115(3):290-6. doi: 10.1038/bjc.2016.209. Epub 2016 Jul 12. PMID 27404453